CLINICAL TRIAL: NCT01955655
Title: Recurrent Crying Spells in Cerebral Palsy With Spastic Quadriparesis - A Crossover Study
Brief Title: Recurrent Crying Spells in Cerebral Palsy
Acronym: RCSCPSQ
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sathbhavana Brain Clinic (Other)
Responsible Party: Principal Investigator, Dr.Nagabhushana Rao Potharaju, Principal Investigator, Sathbhavana Brain Clinic
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RCSCPSQ
Record Dates: First submitted 2013-09-21; First posted 2013-10-07 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: Recurrent Crying Spells
Keywords: Baclofen; cerebral palsy; colic; crying infant; recurrent crying spells; spasticity; therapy
MeSH Terms: conditions — Cerebral Palsy; Colic; Muscle Spasticity | interventions — Baclofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Baclofen (Active Comparator): The starting dose was 0.75 mg/kg in four divided doses daily and was cautiously increased at three-day intervals until crying subsided or symptoms of over dosage or side effects appeared. The usual maximum dose was two mg/kg in four divided doses daily.
  Interventions: Drug: Baclofen
- placebo (Placebo Comparator): Placebo contained fructose powder in equal quantity in packets mimicking those of Baclofen.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Baclofen — Since the therapeutic window of Baclofen is narrow, the lowest dose compatible with an optimal response was used.
  Arms: Baclofen
Other: Placebo
  Other Names: Fructose powder.
  Arms: placebo

SUMMARY:
This is a study of recurrent crying spells in Spastic Cerebral Palsy patients and their treatment.

DETAILED DESCRIPTION:
This is the first study of recurrent crying spells in Cerebral Palsy with Spastic quadriparesis depicting the diagnostic criteria and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent Crying Spells in Cerebral Palsy with Spastic Quadriparesis.
* Age range 0-12 years.

Exclusion Criteria:

* Crying due to known causes (like hunger, sleep, food intolerance etc.),
* Crying that responded to routine management (changes in food or feeding techniques, anticolic, analgesics),
* Fever of ≥100.4ºF (38ºC),
* The infant refuses to eat or drink for more than a few hours, vomits excessively, has bloody stools, or has a change in behavior (lethargy or decreased responsiveness).
* Colic
* Worst ever crying occurring for the first time
* Respiratory, renal and hepatic diseases,
* Progressive encephalopathies,
* Received Baclofen in the previous 30 days

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2005-12; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline cry duration in seconds over a 10-day period while on placebo. | 11th to 20th day and 51st day to 60th day
  Cry duration in seconds over a 10-day period while on placebo was compared to that of Baclofen.

CONTACTS AND LOCATIONS:
Overall Officials: Nagabhushana Rao Potharaju, BScDCHMDDM, Principal Investigator — Sathbhavana Brain Clinic, Secunderabad, India
Locations (1):
- Sathbhavana Brain Clinic, Secunderabad, Andhra Pradesh, India